CLINICAL TRIAL: NCT02158377
Title: A Randomized Controlled Multicenter Study of Trabecular Metal Dental Implants vs.Tapered Screw-Vent Dental Implants Loaded Early vs. Conventionally in the Maxilla and Mandible.
Brief Title: TM vs TSV Implants Loaded Early vs Conventional in Anterior and Posterior Areas
Acronym: TMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSU2011-08D
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: Dental implants; Trabecular Metal dental implants; TSV dental implants; Zimmer Dental; Implant stability; Implant stability quotient (ISQ); Resonance Frequency Analysis (RFA)
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapered Screw-vent implants (TSV) (Active Comparator): TSV implants to replace missing tooth/teeth
  Interventions: Device: Tapered screw-vent implants (TSV)
- Trabecular Metal dental implants (TM) (Experimental): TM dental implants to replace missing tooth/teeth
  Interventions: Device: Trabecular metal dental implants (TM)

INTERVENTIONS:
Device: Trabecular metal dental implants (TM) — Patients receive TM dental implants in this arm. The early stability is measured and compared to the stability of the TSV implants. The implants are loaded and provisionalized early at 3 or 6 weeks if stability permits.
  Arms: Trabecular Metal dental implants (TM)
Device: Tapered screw-vent implants (TSV) — Patients receive TSV dental implants in this arm. The early stability is measured and compared to the stability of the TM implants. The implants are loaded and provisionalized early at 3 or 6 weeks if stability permits.
  Arms: Tapered Screw-vent implants (TSV)

SUMMARY:
Randomized-controlled, multicenter study of Trabecular Metal (TM) and Tapered Screw-Vent (TSV) dental implants loaded early in maxillary and mandibular sites.

DETAILED DESCRIPTION:
This is a randomized, controlled, multicenter study to assess and compare implant stability of Trabecular Metal (TM) dental implants and Tapered Screw-Vent (TSV) implants during the early stages of healing i.e. 21 +/- 2 days and 42+/- 2 days, as well as their short term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Benefit from the implant and restoration
2. Provide a voluntarily signed Informed Consent
3. Must be 18 years or older
4. Have one or more edentulous area(s) in the posterior maxilla or mandible designated for an implant supported restoration
5. The implantation site must have a functional antagonist to obtain full occlusion.
6. Implants adjacent to planned site of implantation should have been in function for at least 1 year.
7. The site intended for implant placement should have healed for at least 4 months from the time of extraction or at least 6 months from any other bone augmentation procedures.
8. The site intended for implant placement should have adequate bone volume to support an implant without the need for augmentation except for minor dehiscence (limited to a vertical height of 2mm), which can be augmented with autogenous bone chips to improve soft tissue attachment.
9. The site intended for implant placement should have residual facial and palatal/lingual plates to be at least 1.0mm thick after implant placement.
10. The site intended for implant placement should have vertical bone volume to extend at least 2.0mm apical to the implant after implant placement.

Exclusion Criteria:

1. Subjects mentally incompetent or unable to understand and provide an Informed Consent
2. Smokers, alcoholics or drug abusers
3. Subjects with systemic conditions such as uncontrolled diabetes, endocrine disorders, heart disease, immune-compromised subjects or mental disorders
4. Use of concurrent medication which inhibits bone metabolism like bisphosphonates, corticosteroids or methotrexate
5. Bleeding disorders and/or anticoagulant therapy
6. Pregnancy
7. Known sensitivity or allergy to any of the implant materials
8. Subjects with bruxism or clenching habits
9. Uncontrolled periodontal or oral pathologies (e.g. mucosal disease, oral lesions)
10. Inadequate oral hygiene
11. History of radiation at the site intended for study implant placement
12. Subjects who have previously failed dental implants at the site intended for study implant placement
13. Subjects participating in another clinical study
14. Subjects who need other surgeries in a site adjacent to the study implant(s)
15. Subjects who need other surgeries in a site non-adjacent to the study implant(s) within 6 months of study implant placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Implant Stability | 3-18 weeks
  Measure of Implant Stability Quotient immediately post implantation

SECONDARY OUTCOMES:
Marginal bone level change | 2 years
  Measurement of bone level surrounding implant

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Wagner, Principal Investigator — Universitatsbedizin Mainz
Locations (3):
- Germany (3):
  - Universitat Regensburg, Regensburg, Bavaria
  - Heinrich Heine Universitat Dusseldorf, Düsseldorf, Nordhein-Westfalen
  - Universitatsmedizin Mainz, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No